CLINICAL TRIAL: NCT02174848
Title: Long-term Safety and Efficacy Study of Deferiprone in Patients With Pantothenate Kinase-Associated Neurodegeneration (PKAN)
Brief Title: Long-term Deferiprone Treatment in Patients With Pantothenate Kinase-Associated Neurodegeneration
Acronym: TIRCON-EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Organization: Chiesi Canada Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIRCON2012V1-EXT; 2012-000845-11 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-26 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pantothenate Kinase-Associated Neurodegeneration
Keywords: Pantothenate Kinase-Associated Neurodegeneration; PKAN; Neurodegeneration with Brain Iron Accumulation; NBIA; Deferiprone; Ferriprox
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration | interventions — Deferiprone; Isoflurophate

STUDY DESIGN:
Intervention Model Description: All participants in this study received the same intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deferiprone (Experimental): All patients will receive deferiprone oral solution.
  Interventions: Drug: Deferiprone oral solution

INTERVENTIONS:
Drug: Deferiprone oral solution — Deferiprone oral solution at a dosage of up to 15 mg per kilogram of body weight, twice a day
  Other Names: DFP

SUMMARY:
Patients with PKAN will be treated with the iron chelator deferiprone for 18 months. Only patients who have completed the earlier study TIRCON2012V1 (NCT01741532), a double-blind placebo-controlled trial in which participants were randomized to receive either deferiprone or placebo for 18 months, are eligible to enroll.

DETAILED DESCRIPTION:
TIRCON2012V1-EXT is a multi-center, single-arm, open-label study. All patients who completed the earlier study TIRCON2012V1 (NCT01741532) are eligible to take part. In the initial study, patients were randomized in a 2:1 ratio to receive 18 months of treatment with either the iron chelator deferiprone or placebo, respectively. In this extension study, all participants will receive deferiprone for 18 months. Thus, depending on which product was received earlier, patients will be on deferiprone for a total of either 1.5 years or 3 years. As in the earlier study, assessments will be carried out every six months to look at the safety of the drug and to see if patients are showing any improvement in dystonia and other symptoms of PKAN.

ELIGIBILITY:
Inclusion Criteria:

* Completed study TIRCON2012V1

Exclusion Criteria:

* Withdrew from the study TIRCON2012V1 for reasons of safety
* Plan to participate in another clinical trial at any time from the day of enrolment until 30 days post-treatment in the current study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Thomas Klopstock, MD, Principal Investigator — Klinikum der Universität München; Nardo Nardocci, MD, Principal Investigator — Foundation Neurological Institute C. Besta; Patrick Chinnery, MD, Principal Investigator — Newcastle University Institute of Human Genetics
Locations (4):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States
- Klinikum der Universität München, Munich, Germany
- Foundation Neurological Institute C. Besta, Milan, Italy
- Newcastle University Institute of Human Genetics, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-DFP: Patients in this group had been randomized to placebo treatment in the TIRCON2012V1 study and were then switched to deferiprone in the extension study. Accordingly, they received up to 18 months of deferiprone treatment over the duration of the two studies.
- DFP-DFP: Patients in this group had been randomized to deferiprone treatment in the TIRCON2012V1 study and then continued on deferiprone in the extension study. Accordingly, they received up to 36 months of deferiprone treatment over the duration of the two studies.
Period: Overall Study
Arm/Group | Placebo-DFP | DFP-DFP
Started | 24 | 44
Provided Post-baseline Efficacy Data | 19 | 43
Completed | 17 | 38
Not Completed | 7 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Worsening of disease | 1 | 1
Not completed — Unable to comply with study requirements | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo-DFP: Patients who received 18 months of placebo treatment in the TIRCON2012V1 study and were then switched to deferiprone in the extension study, so received up to 18 months of deferiprone treatment.
- DFP-DFP: Patients who received 18 months of deferiprone treatment in the TIRCON2012V1 study and continued to receive it in the extension study, so received up to 36 months of deferiprone treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo-DFP | DFP-DFP | Total
Number analyzed (Participants) | 24 | 44 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (13.0) | 22.4 (9.6) | 21.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 10 | 28 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 41 | 63
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
BAD score at baseline [Mean (Standard Deviation); unit: units on a scale] — Scores on the Barry-Albright Dystonia (BAD) scale at baseline of the initial study, prior to the start of treatment, and at baseline of the extension study, following 18 months of treatment with either placebo or deferiprone. Scores on the scale range from 0 to 32, with higher scores indicating more severe dystonia. Population: The baseline efficacy measurements are provided only for the 62 patients who provided at least one post-baseline efficacy assessment and were included in the efficacy analyses of the extension study.
  units on a scale
    BAD score at baseline of initial study: number analyzed (Participants) | 19 | 43 | 62
    BAD score at baseline of initial study | 16.0 (8.0) | 19.4 (8.1) | 18.3 (8.2)
    BAD score at baseline of extension study: number analyzed (Participants) | 19 | 43 | 62
    BAD score at baseline of extension study | 20.4 (8.2) | 21.3 (7.6) | 21.0 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety and tolerability were assessed based on changes in: frequency of adverse events (AEs), frequency of serious adverse events (SAEs), and discontinuation due to AEs. No statistical comparison between the groups was conducted as all participants received the same study product.
Time Frame: 18 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo-DFP: Patients in this group had been randomized to placebo treatment in the TIRCON2012V1 study and were then switched to deferiprone in the extension study. Accordingly, they received up to 18 months of deferiprone treatment.
- DFP-DFP: Patients in this group had been randomized to deferiprone treatment in the TIRCON2012V1 study and then continued on deferiprone in the extension study. Accordingly, they received up to 36 months of deferiprone treatment.
Arm/Group | Placebo-DFP | DFP-DFP
Number analyzed (Participants) | 24 | 44
Participants
  Number of patients with at least one AE | 22 | 42
  Number of patients with at least one SAE | 12 | 14
  Number of patients who withdrew due to an AE | 2 | 1

2. Secondary Outcome: Change in Score on the BAD Scale -- Comparison of Treatment Groups Over Each Study
Description: The Barry-Albright Dystonia (BAD) scale is an instrument for rating the severity of dystonia in eight body regions. The individual scores are summed to provide a total score that ranges from 0 to 32; the higher the score, the more severe the dystonia. Patients were assessed for the change in total BAD score over the course of both the initial study (during which one group received placebo and the other received deferiprone) and the extension study (during which both groups received deferiprone).
Time Frame: Baseline and Month 18 of each study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-DFP | DFP-DFP
Number analyzed (Participants) | 19 | 43
score on a scale
  Change in BAD score over initial study | 4.4 (4.8) | 1.9 (3.2)
  Change in BAD score over extension study | 1.4 (3.7) | 1.4 (2.4)
Statistical Analysis 1: Comparison: Placebo-DFP vs DFP-DFP; This comparison is for the initial study, during which patients in the placebo-DFP group received placebo and patients in the DFP-DFP group received deferiprone; Test type: Superiority; p = 0.0500, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo-DFP vs DFP-DFP; This comparison is for the extension study, during which patients in both groups received deferiprone; Test type: Superiority; p = 0.9781, t-test, 2 sided

3. Secondary Outcome: Change in Score on the BAD Scale -- Comparison of Placebo-DFP Patients Across Studies
Description: The Barry-Albright Dystonia (BAD) scale is an instrument for rating the severity of dystonia in eight body regions. The individual scores are summed to provide a total score that ranges from 0 to 32; the higher the score, the more severe the dystonia. Patients were assessed for the change in total BAD score over the course of each study.
Time Frame: Baseline and Month 18 of each study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo-DFP in Initial Study: During the initial study, patients in the placebo-DFP group received 18 months of treatment with placebo
- Placebo-DFP in Extension Study: During the extension study, patients in the placebo-DFP group received up to 18 months of treatment with deferiprone
Arm/Group | Placebo-DFP in Initial Study | Placebo-DFP in Extension Study
Number analyzed (Participants) | 19 | 19
score on a scale | 4.4 (4.8) | 1.4 (3.7)
Statistical Analysis 1: Comparison: Placebo-DFP in Initial Study vs Placebo-DFP in Extension Study; Test type: Superiority; p = 0.0206, paired t-test

4. Secondary Outcome: Change in Score on the BAD Scale -- Comparison of DFP-DFP Patients Across Studies
Description: The Barry-Albright Dystonia (BAD) scale is an instrument for rating the severity of dystonia in eight body regions. The individual scores are summed to provide a total score that ranges from 0 to 32; the higher the score, the more severe the dystonia. Patients were assessed for the change in total BAD score over the course of the study.
Time Frame: Baseline and Month 18 of each study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DFP-DFP Group in Initial Study: During the initial study, patients in the DFP-DFP group received 18 months of treatment with deferiprone
- DFP-DFP Group in Extension Study: During the extension study, patients in the DFP-DFP group received up to an additional 18 months of treatment with deferiprone
Arm/Group | DFP-DFP Group in Initial Study | DFP-DFP Group in Extension Study
Number analyzed (Participants) | 43 | 43
score on a scale | 1.9 (3.2) | 1.4 (2.4)
Statistical Analysis 1: Comparison: DFP-DFP Group in Initial Study vs DFP-DFP Group in Extension Study; Test type: Superiority; p = 0.2684, paired t-test

5. Secondary Outcome: Proportion of Patients With Improved or Unchanged BAD Score
Description: Patients were deemed to be responders if their BAD total score either improved or remained unchanged from baseline, with baseline being the start of each study for the placebo-DFP group and the start of the initial study for the DFP-DFP group
Time Frame: Month 18 of each study
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-DFP | DFP-DFP
Number analyzed (Participants) | 19 | 43
Participants
  Completion of initial study | 3 | 17
  Completion of 18 months of deferiprone treatment | 9 | 17
Statistical Analysis 1: Comparison: Placebo-DFP vs DFP-DFP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0821, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo-DFP vs DFP-DFP; For the placebo-DFP group, the comparison is of the scores at the start vs. the end of the extension study; for the DFP-DFP group, the comparison is of the scores at the start vs. the end of the initial study; Test type: Superiority; p = 0.5885, t-test, 2 sided

6. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Comparison of Placebo-DFP Patients Across Studies
Description: The Patient Global Impression of Improvement (PGI-I) is a global index used to rate the response of a condition to a therapy. Patients were asked at each post-baseline visit to rate their overall condition since the start of the extension study on a 7-point rating scale: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Month 18 of each study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-DFP in Initial Study | Placebo-DFP in Extension Study
Number analyzed (Participants) | 19 | 19
score on a scale | 4.4 (1.5) | 4.7 (1.4)
Statistical Analysis 1: Comparison: Placebo-DFP in Initial Study vs Placebo-DFP in Extension Study; Test type: Superiority; p = 0.3306, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Safety data were collected from the time of first dose until the end of the study (up to 18 months)
Groups:
- All Patients: All participants received deferiprone during the extension study
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 2/68
Serious Adverse Events (participants affected / at risk) | 33/68
Other Adverse Events (participants affected / at risk) | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=68)
Neutropenia (Blood and lymphatic system disorders) | 4 (7)
Cyanosis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Medical device site inflammation (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Obstruction (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Bacterial disease carrier (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Infective glossitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Chemical eye injury (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Device function test (Investigations) | 1 (1)
Physical examination (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dystonia (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 1 (1)
Hyporesponsive to stimuli (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Device stimulation issue (Product Issues) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 1 (1)
Dental operation (Surgical and medical procedures) | 1 (1)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 4 (4)
Hip surgery (Surgical and medical procedures) | 1 (1)
Intrathecal pump insertion (Surgical and medical procedures) | 1 (1)
Jejunostomy (Surgical and medical procedures) | 1 (1)
Medical device battery replacement (Surgical and medical procedures) | 2 (2)
Medical device change (Surgical and medical procedures) | 2 (2)
Medical device implantation (Surgical and medical procedures) | 3 (3)
Medical device removal (Surgical and medical procedures) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (5)
Tracheostomy tube removal (Surgical and medical procedures) | 1 (1)
Wound treatment (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=68)
Anemias (Blood and lymphatic system disorders) | 12 (27)
Abdominal pain upper (Gastrointestinal disorders) | 8 (16)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 10 (13)
Condition aggravated (General disorders) | 17 (25)
Pain (General disorders) | 5 (5)
Pyrexia (General disorders) | 20 (64)
Bronchitis (Infections and infestations) | 6 (30)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (22)
Upper respiratory tract infection (Infections and infestations) | 13 (19)
Urinary tract infection (Infections and infestations) | 6 (8)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Laceration (Injury, poisoning and procedural complications) | 8 (20)
Body temperature increased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 10 (26)
Serum ferritin decreased (Investigations) | 18 (25)
Iron deficiency (Metabolism and nutrition disorders) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (11)
Pain in extremity (Metabolism and nutrition disorders) | 14 (26)
Aphasia (Nervous system disorders) | 5 (6)
Ataxia (Nervous system disorders) | 4 (4)
Balance disorder (Nervous system disorders) | 5 (5)
Dystonia (Nervous system disorders) | 32 (74)
Headache (Nervous system disorders) | 19 (64)
Somnolence (Nervous system disorders) | 6 (8)
Tremor (Nervous system disorders) | 4 (7)
Agitation (Psychiatric disorders) | 5 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retained title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the trial. Such publications shall not be made without the prior written consent of Sponsor. Neither Party will use the other Party's name in connection with any publication or promotion without the other Party's prior written consent. However, Sponsor has the right to publish appropriate information in order to satisfy regulatory requirements.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT02174848/SAP_000.pdf
  • Study Protocol (2014-08-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT02174848/Prot_001.pdf